CLINICAL TRIAL: NCT00519467
Title: An Open, Randomised, Multi-centre Dose Ranging Phase II Study to Evaluate LAPDAP in Combination With Three Different Doses of Artesunate
Brief Title: Safety and Efficacy Dose of Artesunate Used in Combination With LAPDAP Treatment of Uncomplicated Falciparum Malaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SB-714703/003
Record Dates: First submitted 2007-08-20; First posted 2007-08-22 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Malaria
Keywords: dose-ranging study; SB-714703; artesunate,; malaria; CDA,; chlorproguanil,; dapsone,
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Chlorproguanil-dapsone-artesunate (CDA)

SUMMARY:
Drug resistance to a range of antimalarial treatments has become widespread in Africa, South East Asia and South America. Because the rapid spread of drug resistance threatens a public health disaster in these areas of the world and to comply with the WHO-Roll Back Malaria policy of using Artemisinin-based combination therapies (ACT), there is a need to develop new, safe, effective and affordable ACT.

Chlorproguanil-dapsone-artesunate (CDA)is a new ACT that is being developed for the treatment of uncomplicated falciparum malaria in Africa.

ELIGIBILITY:
Inclusion Criteria:

* Presentation to a healthcare facility with probable uncomplicated clinical malaria
* Adults aged between 18 and 60 years , or children aged between 12 and 120 months
* Weight between 5 and 85kg
* Pure [on microscopic grounds] screening P. falciparum parasitaemia in children from 25,000 to 100,000ul-1, or in adults from 10,000 to 100,000ul-1. [The parasitaemia range for adults was originally set at 25,000 to 100,000µl-1 and changed to 10,000 to 100,000µl-1 in protocol amendment 3 dated 05 May 2004]
* Written or oral witnessed consent obtained from subject, parent or guardian
* Compliance with the requirements of the protocol which include a hospital stay of 4 days and 3 nights and regular blood samples by finger-prick (children) or via a cannula (adults)
* A negative pregnancy test for women of child-bearing age on enrolment

Exclusion Criteria:

* Features of severe/complicated falciparum malaria
* Known allergy to sulphonamides
* Evidence of any concomitant infection at the time of presentation (including P. ovale and P. malaria)
* Any other underlying disease that would compromise the diagnosis and the evaluation of the response to the study medication (including clinical symptoms of immunosuppression, tuberculosis and bacterial infection)
* Treatment in the 28-days prior to screening with sulfadoxine/pyrimethamine (FANSIDAR, CELOXINE), sulfalene/pyrimethamine (METAKELFIN), mefloquine-sulfadoxinepyrimethamine (FANSIMET), chloroquine* (NIVAQUINE); treatment in the 21-days prior to screening with mefloquine, or 7-days prior to screening with amodiaquine, halofantrine, quinine (full course), atovaquone - proguanil, artemisinins, co-artemether, tetracycline or clindamycin, or treatment for 5 half-lives prior to screening with drugs that have a potential anti-malarial activity (e.g. co-trimoxazole in the previous 60 hours)
* Use of an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to screening
* Previous participation in this study
* A positive pregnancy test at enrolment, women of child-bearing age who do not take a pregnancy test or female subjects who are breast-feeding an infant for the duration of the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2003-06; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Treatment differences between 1,2, or 4mg/kg artesunate with a fixed dose of Chlorproguanil-dapsone (LAPDAP), as measured by determination of PC90 (time to achieve reduction of parasitaemia by 90% of baseline)

SECONDARY OUTCOMES:
The key secondary efficacy endpoint is parasite viability (the proportion of ring-form parasites developing to schizonts) determined from rich adult data and confirmed with more sparse child data

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Blantyre, Malawi
- GSK Investigational Site, Banjul, The Gambia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Miller AK, Bandyopadhyay N, Wootton DG, Duparc S, Kirby PL, Winstanley PA, Ward SA. Pharmacokinetics of chlorproguanil, dapsone, artesunate and their major metabolites in patients during treatment of acute uncomplicated Plasmodium falciparum malaria. Eur J Clin Pharmacol. 2009 Oct;65(10):977-87. doi: 10.1007/s00228-009-0672-1. Epub 2009 Jun 11. PMID 19517101
- [Derived] Wootton DG, Opara H, Biagini GA, Kanjala MK, Duparc S, Kirby PL, Woessner M, Neate C, Nyirenda M, Blencowe H, Dube-Mbeye Q, Kanyok T, Ward S, Molyneux M, Dunyo S, Winstanley PA. Open-label comparative clinical study of chlorproguanil-dapsone fixed dose combination (Lapdap) alone or with three different doses of artesunate for uncomplicated Plasmodium falciparum malaria. PLoS One. 2008 Mar 5;3(3):e1779. doi: 10.1371/journal.pone.0001779. PMID 18320064
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 714703/003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 714703/003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 714703/003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 714703/003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 714703/003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 714703/003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 714703/003 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register